CLINICAL TRIAL: NCT02051335
Title: A Randomized, Double-Blind, Placebo Controlled, 4-Period, Cross-Over Study to Evaluate the Effects of Single Oral Administrations of Roflumilast in Combination With Donepezil on Reversing Scopolamine (Hyoscine) Induced Deficits in Psychomotor and Cognitive Function in Healthy Adults
Brief Title: Roflumilast and Donepezil to Reverse Scopolamine Induced Cognitive Deficits in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROF-ALZ_102; 2012-002089-11 (EudraCT Number); U1111-1151-7178 (Registry Identifier: UTN (WHO))
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-09

CONDITIONS: Memory Impairment; Alzheimer's Disease
Keywords: Drug therapy
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease | interventions — Roflumilast; Donepezil; Scopolamine; Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (ABDC) (Experimental): Roflumilast placebo-matching tablets, orally, donepezil placebo-matching overencapsulated tablets, orally, and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 1, followed by roflumilast placebo-matching tablets, orally, donepezil 10 mg, overencapsulated tablets, orally and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 2, followed by roflumilast Dose A tablets, orally, donepezil 10 mg, overencapsulated tablets, orally and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 3, followed by roflumilast Dose A tablets, orally, donepezil placebo-matching overencapsulated tablets, orally, and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 4. Each treatment period is separated by a 14-day washout period.
  Interventions: Drug: Roflumilast; Drug: Roflumilast placebo; Drug: Donepezil; Drug: Donepezil placebo; Drug: Scopolamine
- Sequence 2 (BCAD) (Experimental): Roflumilast placebo-matching tablets, orally, donepezil 10 mg, overencapsulated tablets, orally and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 1, followed by roflumilast Dose A tablets, orally, donepezil placebo-matching overencapsulated tablets, orally, and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 2, followed by roflumilast placebo-matching tablets, orally, donepezil placebo-matching overencapsulated tablets, orally, and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 3, followed by roflumilast Dose A tablets, orally, donepezil 10 mg, overencapsulated tablets, orally and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 4. Each treatment period is separated by a 14-day washout period.
  Interventions: Drug: Roflumilast; Drug: Roflumilast placebo; Drug: Donepezil; Drug: Donepezil placebo; Drug: Scopolamine
- Sequence 3 (CDBA) (Experimental): Roflumilast Dose A tablets, orally, donepezil placebo-matching overencapsulated tablets, orally, and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 1, followed by roflumilast Dose A tablets, orally, donepezil 10 mg, overencapsulated tablets, orally and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 2, followed by roflumilast placebo-matching tablets, orally, donepezil 10 mg, overencapsulated tablets, orally and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 3, followed by roflumilast placebo-matching tablets, orally, donepezil placebo-matching overencapsulated tablets, orally, and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 4. Each treatment period is separated by a 14-day washout period.
  Interventions: Drug: Roflumilast; Drug: Roflumilast placebo; Drug: Donepezil; Drug: Donepezil placebo; Drug: Scopolamine
- Sequence 4 (DACB) (Experimental): Roflumilast Dose A tablets, orally, donepezil 10 mg, overencapsulated tablets, orally and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 1, followed by roflumilast placebo-matching tablets, orally, donepezil placebo-matching overencapsulated tablets, orally, and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 2, followed by roflumilast Dose A tablets, orally, donepezil placebo-matching overencapsulated tablets, orally, and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 3, followed by roflumilast placebo-matching tablets, orally, donepezil 10 mg, overencapsulated tablets, orally and scopolamine 0.5 mg subcutaneous injection, once, Day 1, Period 4. Each treatment period is separated by a 14-day washout period.
  Interventions: Drug: Roflumilast; Drug: Roflumilast placebo; Drug: Donepezil; Drug: Donepezil placebo; Drug: Scopolamine

INTERVENTIONS:
Drug: Roflumilast — Roflumilast tablets
  Other Names: Daxas
Drug: Roflumilast placebo — Roflumilast placebo-matching tablets
Drug: Donepezil — Donepezil overencapsulated tablets
  Other Names: Aricept
Drug: Donepezil placebo — Donepezil placebo-matching overencapsulated tablets
Drug: Scopolamine — Scopolamine subcutaneous injection
  Other Names: Hyoscine hydrobromide

SUMMARY:
The purpose of this study is to determine whether scopolamine-induced cognitive impairment is attenuated by the administration of roflumilast in combination with donepezil.

DETAILED DESCRIPTION:
The drug being tested in this study is called roflumilast. Roflumilast is being tested as a potential treatment for Alzheimer's disease. This study will look at roflumilast combined with a medication called donepezil, and their ability to reverse mimicked Alzheimer's disease symptoms that have been brought on by administration of a drug called scopolamine.

The study will enroll up to 28 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of four treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need). All participants will receive the following treatments at varying time points throughout the study:

* Roflumilast Dose A tablets
* Donepezil 10 mg capsules
* Placebo (dummy inactive pill) - this is a tablet or capsule that looks like the study drug but has no active ingredient
* Scopolamine 0.5 mg subcutaneous injection.

All participants will be asked to take 2 tablets and 1 capsule and will receive a scopolamine subcutaneous injection on the first day of 4 separate study periods. Participants will then be assessed for how the scopolamine affects their mental processes and whether the study drug improves this.

This single-center trial will be conducted in England. The overall time to participate in this study is up to 95 days. Participants will make 7 visits to the clinic, including 4 separate periods of 2 days confinement to the clinic, and a follow-up assessment 14 days after the last treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is a healthy adult male.
4. Is aged 18 to 45 years, inclusive, at the time of informed consent.
5. Weighs at least 60 kg and has a body mass index (BMI) between 18 and 32 kg/m^2 inclusive at Screening.
6. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
7. Has clinical laboratory evaluations (including clinical chemistry, hematology and complete urinalysis) within the reference range for the testing laboratory, unless the results are deemed not to be clinically significant (CS) by the investigator at screening and Day -1 (Check-in) of Period 1.

Exclusion Criteria:

1. Has received any investigational compound within 3 months prior to the first dose of study medication.
2. Has received roflumilast, donepezil, or scopolamine in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality which may impact the ability of the participant to participate or potentially confound the study results.
5. Contraindications to scopolamine: hypersensitivity to scopolamine and other belladonna alkaloids, and/or any component of the formulation, serious allergic reactions, wide and narrow angle glaucoma, gastrointestinal motility disorders (such as constipation, gastroesophageal reflux disease, irritable bowel syndrome), benign prostatic hyperplasia with urinary retention, asthma, chronic obstructive pulmonary disease (COPD), seizures, coronary artery disease, hypertension, and congestive heart failure.
6. Participants with existing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder according to the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, as assessed by the Mini International Neuropsychiatric Interview (MINI) or acute psychiatric episode within 6 months of Screening.
7. Has a known hypersensitivity to any component of the formulation of roflumilast, donepezil, scopolamine, or related compounds.
8. Has a positive urine drug result for drugs of abuse at Screening or Day -1 (Check-in) of each Period.
9. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the screening visit or is unwilling to agree to abstain from drug use or excessive alcohol use throughout the study.
10. Has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products.
11. Intends to donate sperm during the course of this study or for 12 weeks thereafter.
12. Any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking roflumilast, donepezil, scopolamine, or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
13. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, or erosive esophagitis, frequent [more than once per week] occurrence of heartburn.
14. Has had any surgical intervention within 6 months that may impact the bioavailability of the compound (eg, cholecystectomy, bariatric surgery).
15. Has a history of cancer within the past 5 years prior to the first dose of study medication. This criterion does not include those participants with basal cell or stage I squamous cell carcinoma of the skin who are eligible.
16. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), human immunodeficiency virus (HIV) antibody/antigen at Screening.
17. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in on Day -1 (Check-in of Period 1).
18. Cotinine test is positive at Screening or Check-in (Day -1 of each Period).
19. Has poor peripheral venous access.
20. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 3 months prior to Day 1 of Period 1.
21. Has a Screening or Day -1 (Check-in) of Period 1 abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator or qualified delegate.
22. Has abnormal Screening or Day -1 (Check-in) of Period 1 laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 the upper limits of normal.
23. Has a current diagnosis or history of glaucoma or had a first-degree relative diagnosed with glaucoma.
24. Has a risk of suicide according to the investigator's clinical judgment (eg, per Columbia-Suicide Severity Rating Scale (C-SSRS) or has made a suicide attempt in the previous 6 months).
25. Has a history of depression associated with suicidal thinking and/or behavior.
26. 26. In the opinion of the investigator or sponsor, the participant is unsuitable for inclusion in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United Kingdom from 16 January 2014 to 17 May 2014.
Pre-assignment Details: Participants with a diagnosis of Alzeimer's disease were enrolled equally in a 4 period, 4 treatment crossover study. Treatment A: Placebo, Treatment B: Donepezil, Treatment C: Roflumilast and Treatment D: Roflumilast + Donepezil. All participants received scopolamine on Day 1 of each treatment period.
Period: Period 1
Arm/Group | Sequence 1 (ABDC) | Sequence 2 (BCAD) | Sequence 3 (CDBA) | Sequence 4 (DACB)
Started | 7 | 7 | 7 | 6
Completed | 7 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 (ABDC) | Sequence 2 (BCAD) | Sequence 3 (CDBA) | Sequence 4 (DACB)
Started | 7 | 7 | 7 | 4 (2 Participants received treatment in Period 1 but discontinued prior to Period 2.)
Completed | 7 | 7 | 7 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 (ABDC) | Sequence 2 (BCAD) | Sequence 3 (CDBA) | Sequence 4 (DACB)
Started | 7 | 7 | 5 (2 Participants received treatment in Period 2 but discontinued prior to Period 3.) | 4
Completed | 7 | 7 | 5 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 (ABDC) | Sequence 2 (BCAD) | Sequence 3 (CDBA) | Sequence 4 (DACB)
Started | 7 | 7 | 5 | 4
Completed | 7 | 7 | 5 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 (ABDC) | Sequence 2 (BCAD) | Sequence 3 (CDBA) | Sequence 4 (DACB) | Total
Number analyzed (Participants) | 7 | 7 | 7 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (7.69) | 28.4 (6.73) | 34.1 (6.89) | 29.8 (5.12) | 31.1 (6.71)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 7 | 7 | 6 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 2 | 0 | 1 | 6
  Black or African American | 0 | 1 | 3 | 2 | 6
  White | 4 | 4 | 4 | 3 | 15
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7 | 7 | 7 | 6 | 27
Height [Mean (Standard Deviation); unit: cm] | 178.7 (6.65) | 177.3 (6.87) | 179.0 (5.23) | 174.5 (5.79) | 177.5 (6.08)
Weight [Mean (Standard Deviation); unit: kg] | 82.16 (9.759) | 78.61 (7.189) | 81.53 (4.476) | 75.05 (7.036) | 79.50 (7.473)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.76 (3.173) | 25.09 (2.683) | 25.49 (1.670) | 24.68 (2.568) | 25.27 (2.462)
Smoking Classification [Number; unit: participants]
  Never Smoked | 7 | 7 | 6 | 6 | 26
  Current Smoker | 0 | 0 | 0 | 0 | 0
  Ex-smoker | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Verbal Recall Memory (VRM) Total Number of Correct Responses for Delayed Recall at 1 Hour After Scopolamine Administration
Description: VRM measures the ability to encode and subsequently retrieve verbal information. This task begins with the first presentation phase in which 18 words are shown in turn on the screen. The participant is then asked to recall as many words as possible during the first immediate recall phase. The same 18 words are then shown in a second presentation phase which is followed by a second immediate recall phase. After a delay of approximately 20-30 minutes, a delayed recall stage is completed. The possible range of correct responses is 0 (worst) to 18 (best). Higher number of correct responses in the test indicates a better outcome. A negative change from baseline indicates a worsening of the score.
Time Frame: Baseline and 1 hour after scopolamine administration on Day 1 of each treatment period. Baseline is defined as the assessment 1 hour before roflumilast/donepezil administration (3 hours before scopolamine administration).
Population: Participants from the Full Analysis Set with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: correct responses
Groups:
- A: Placebo: Roflumilast placebo-matching tablets, orally, donepezil placebo-matching overencapsulated tablets, orally, and scopolamine 0.5 mg subcutaneous injection, once, Day 1 in any of the 4 treatment periods.
- B: Donepezil 10 mg: Roflumilast placebo-matching tablets, orally, donepezil 10 mg, overencapsulated tablets, orally and scopolamine 0.5 mg subcutaneous injection, once, Day 1 in any of the 4 treatment periods.
- C: Roflumilast Dose A: Roflumilast Dose A tablets, orally, donepezil placebo-matching overencapsulated tablets, orally, and scopolamine 0.5 mg subcutaneous injection, once, Day 1 in any of the 4 treatment periods.
- D: Roflumilast Dose A + Donepezil 10 mg: Roflumilast Dose A tablets, orally, donepezil 10 mg, overencapsulated tablets, orally and scopolamine 0.5 mg subcutaneous injection, once, Day 1 in any of the 4 treatment periods.
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Number analyzed (Participants) | 23 | 23 | 25 | 27
correct responses | -6.7 (3.02) | -7.0 (3.33) | -7.4 (3.62) | -6.6 (2.68)
Statistical Analysis 1: Comparison: A: Placebo vs B: Donepezil 10 mg; Test type: Superiority or Other; p = 0.573, ANOVA — P-values were obtained using an ANOVA model with sequence, period, and treatment as fixed effects and participant nested within sequence as a random effect; LS mean difference = -0.31, 95% CI 2-sided [-1.4 to 0.8], Standard Error of Mean 0.556
Statistical Analysis 2: Comparison: A: Placebo vs C: Roflumilast Dose A; Test type: Superiority or Other; p = 0.210, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.70, 95% CI 2-sided [-1.8 to 0.4], Standard Error of Mean 0.550
Statistical Analysis 3: Comparison: A: Placebo vs D: Roflumilast Dose A + Donepezil 10 mg; Test type: Superiority or Other; p = 0.821, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 0.12, 95% CI 2-sided [-1.0 to 1.2], Standard Error of Mean 0.547
Statistical Analysis 4: Comparison: B: Donepezil 10 mg vs D: Roflumilast Dose A + Donepezil 10 mg; Test type: Superiority or Other; p = 0.426, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 0.44, 95% CI 2-sided [-0.7 to 1.5], Standard Error of Mean 0.549
Statistical Analysis 5: Comparison: C: Roflumilast Dose A vs D: Roflumilast Dose A + Donepezil 10 mg; Test type: Superiority or Other; p = 0.126, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 0.82, 95% CI 2-sided [-0.2 to 1.9], Standard Error of Mean 0.530

2. Primary Outcome: Change From Baseline in the Verbal Recall Memory (VRM) Total Number of Correct Responses for Immediate Recall at 1 Hour After Scopolamine Administration
Description: VRM measures the ability to encode and subsequently retrieve verbal information. This task begins with the first presentation phase in which 18 words are shown in turn on the screen. The participant is then asked to recall as many words as possible during the first immediate recall phase. The possible range of correct responses is 0 (worst) to 18 (best). Higher number of correct responses in the test indicates a better outcome. A negative change from baseline indicates a worsening of the score.
Time Frame: Baseline and 1 hour after scopolamine administration on Day 1 of each treatment period.
Population: Participants from the Full Analysis Set with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Number analyzed (Participants) | 23 | 23 | 25 | 27
correct responses | -9.8 (4.77) | -7.7 (4.37) | -10.6 (5.09) | -7.7 (4.42)
Statistical Analysis 1: Comparison: A: Placebo vs B: Donepezil 10 mg; Test type: Superiority or Other; p = 0.057, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 1.93, 95% CI 2-sided [-0.1 to 3.9], Standard Error of Mean 0.992
Statistical Analysis 2: Comparison: A: Placebo vs C: Roflumilast Dose A; Test type: Superiority or Other; p = 0.394, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.84, 95% CI 2-sided [-2.8 to 1.1], Standard Error of Mean 0.981
Statistical Analysis 3: Comparison: A: Placebo vs D: Roflumilast Dose A + Donepezil 10 mg; Test type: Superiority or Other; p = 0.042, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 2.01, 95% CI 2-sided [0.1 to 4.0], Standard Error of Mean 0.972
Statistical Analysis 4: Comparison: B: Donepezil 10 mg vs D: Roflumilast Dose A + Donepezil 10 mg; Test type: Superiority or Other; p = 0.928, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 0.09, 95% CI 2-sided [-1.9 to 2.0], Standard Error of Mean 0.974
Statistical Analysis 5: Comparison: C: Roflumilast Dose A vs D: Roflumilast Dose A + Donepezil 10 mg; Test type: Superiority or Other; p = 0.004, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 2.86, 95% CI 2-sided [1.0 to 4.7], Standard Error of Mean 0.943

3. Secondary Outcome: Change From Baseline in the Verbal Recall Memory (VRM) Total Number of Correct Responses for Immediate and Delayed Recall at 2 and 4 Hours After Scopolamine Administration
Description: as for outcome 1
Time Frame: Baseline and 2 and 4 hours after scopolamine administration on Day 1 of each treatment period.
Population: Participants from the Full Analysis Set with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Number analyzed (Participants) | 23 | 23 | 25 | 27
correct responses
  Immediate Recall: 2 hours post Scopolamine | -10.1 (5.02) | -7.3 (4.06) | -9.9 (5.20) | -6.5 (4.38)
  Immediate Recall: 4 hours post Scopolamine | -8.3 (5.64) | -7.6 (4.59) | -7.9 (4.50) | -6.1 (4.23)
  Delayed Recall: 2 hours post Scopolamine | -6.3 (2.08) | -5.6 (2.87) | -6.8 (3.67) | -5.9 (3.06)
  Delayed Recall: 4 hours post Scopolamine | -5.5 (2.64) | -5.6 (3.34) | -5.9 (2.98) | -5.3 (2.50)

4. Secondary Outcome: Change From Baseline in the Paired Associates Learning (PAL) Total Number of Errors Adjusted at All Time-points Assessed After Scopolamine Administration
Description: PAL assesses visuospatial associative learning and memory. Boxes are displayed on the screen and open in a randomised order to reveal a number of patterns. The patterns are then displayed in the middle of the screen, one at a time, and the participant must touch the box where the pattern was originally located. If the participant makes an error, the patterns are re-presented to remind the participant of their locations. If the participant has not responded correctly within six attempts, ie, one presentation and five re-presentations, the task is terminated. As the task progresses the difficulty level increases with the number of patterns to be remembered. For participants who fail to complete all levels, an adjusted total is calculated that takes into account errors predicted in the stages that were not attempted. The possible range for total errors is 0 (best) to 91 (worst). Fewer number of errors in the test indicates a better outcome.
Time Frame: Baseline and at 1, 2 and 4 hours after scopolamine administration on Day 1 of each treatment period.
Population: Participants from the Full Analysis Set with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Number analyzed (Participants) | 23 | 23 | 25 | 27
errors
  1 hour post Scopolamine | 8.0 (12.73) | 11.5 (15.98) | 1.6 (10.70) | 7.5 (14.38)
  2 hours post Scopolamine | 3.0 (10.11) | 3.0 (7.23) | -0.7 (11.96) | 2.9 (9.12)
  4 hours post Scopolamine | 2.3 (9.09) | 7.7 (16.00) | 0.2 (8.34) | 3.1 (9.31)

5. Secondary Outcome: Change From Baseline in the Rapid Visual Information Processing (RVP) A Prime Signal Detection at All Time-points Assessed After Scopolamine Administration
Description: RVP is a task of continuous performance and visual sustained attention. The task consists of a 2-minute practice stage and a 7-minute assessed stage. There is a white box in the centre of the screen in which single digits from 2 to 9 appear one at a time in a pseudo-random order at a rate of 100 digits per minute. Participants must detect target sequences of digits (2-4-6, 3-5-7, and 4-6-8) and touch a button when they see the last digit of a target sequence. Nine target sequences appear every 100 numbers. A prime (A') is a signal detection measure that reflects target sensitivity regardless of the participant's tendency, or bias, to respond. Detection sensitivity for RVP A' prime: 0 to 1. Lower numbers in the test indicates worsening in the performance.
Time Frame: Baseline and at 1, 2 and 4 hours after scopolamine administration on Day 1 of each treatment period.
Population: Participants from the Full Analysis Set with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Number analyzed (Participants) | 23 | 23 | 25 | 27
unitless
  1 hour post Scopolamine | -0.0184 (0.03206) | -0.0107 (0.03661) | -0.0290 (0.03090) | -0.0157 (0.03742)
  2 hours post Scopolamine | -0.0297 (0.03799) | -0.0151 (0.03249) | -0.0315 (0.03810) | -0.0282 (0.04667)
  4 hours post Scopolamine | -0.0201 (0.03972) | -0.0106 (0.02948) | -0.0227 (0.03534) | -0.0114 (0.03530)

6. Secondary Outcome: Change From Baseline in the Rapid Visual Information Processing (RVP) Median Latency at All Time-points Assessed After Scopolamine Administration
Description: RVP is a task of continuous performance and visual sustained attention. The task consists of a 2-minute practice stage and a 7-minute assessed stage. There is a white box in the centre of the screen in which single digits from 2 to 9 appear one at a time in a pseudo-random order at a rate of 100 digits per minute. Participants must detect target sequences of digits (2-4-6, 3-5-7, and 4-6-8) and touch a button when they see the last digit of a target sequence. Nine target sequences appear every 100 numbers. Assessment will be based on a median latency. The possible range for RVP median latency is 100 (worst) to 1900 (best). Higher number in the test indicates a better outcome. "Median latency" is a measure captured by computerized test measure and given as "one" time value (between 100 and 1900). The "mean" of these values is presented.
Time Frame: Baseline and at 1, 2 and 4 hours after scopolamine administration on Day 1 of each treatment period.
Population: Participants from the Full Analysis Set with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Number analyzed (Participants) | 23 | 23 | 25 | 27
msec
  1 hour post Scopolamine | 10.63 (39.631) | -7.35 (36.659) | 5.62 (36.538) | 2.59 (42.550)
  2 hours post Scopolamine | 10.83 (45.635) | -4.89 (42.713) | 10.62 (40.063) | 0.13 (55.005)
  4 hours post Scopolamine | 13.13 (42.087) | -5.39 (33.696) | 3.90 (39.485) | -8.98 (41.002)

7. Secondary Outcome: Change From Baseline in the Spatial Working Memory (SWM) Total Number of Between Errors at the 10-Box Stage and the 12-Box Stage at All Time-points Assessed After Scopolamine Administration
Description: SWM assesses the ability to retain spatial information and manipulate it in working memory. In this task, colored boxes are shown on the screen, and participants must search for blue tokens by touching the colored boxes to open them. When the blue token has been found the participant has to place the token in the black column ('home') on the right-hand side of the screen by touching this area. The participant must not return to a box where a token has previously been found. The task becomes more difficult as the number of boxes increases (one trial at each of 6-box and 8-box stages; three trials at each of 10-box and 12-box stages). Between Errors is the total number of times the participant revisits a box in which a token has previously been found in the same problem. The possible range of errors is 0 (best) to 1040 (worst). Lower number of errors in the test indicates a better outcome.
Time Frame: Baseline and at 1, 2 and 4 hours after scopolamine administration on Day 1 of each treatment period.
Population: Participants from the Full Analysis Set with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Number analyzed (Participants) | 23 | 23 | 25 | 27
errors
  1 hour post Scopolamine | 23.8 (36.96) | 25.7 (27.77) | 31.7 (22.66) | 16.5 (22.87)
  2 hours post Scopolamine | 28.4 (22.57) | 13.4 (27.47) | 29.6 (23.88) | 18.2 (22.18)
  4 hours post Scopolamine | 31.1 (29.88) | 19.7 (25.46) | 32.8 (26.62) | 7.7 (21.09)

8. Secondary Outcome: Percentage of Participants Who Experience at Least 1 Treatment Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as any adverse event, regardless of relationship to study drug that occurs or worsens after the first dose of study drug and no more than 14 days after the last dose of study drug.
Time Frame: Day 1 up to Day 95
Population: Safety Analysis Set included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Number analyzed (Participants) | 23 | 23 | 25 | 27
percentage of participants | 30.4 | 65.2 | 24.0 | 51.9

9. Secondary Outcome: Percentage of Participants With Markedly Abnormal Safety Laboratory Tests
Description: The percentage of participants with any markedly abnormal standard safety laboratory values, including hematology, serum chemistries, and urinalysis. LLN=lower limit of normal. ULN=upper limit of normal.
Time Frame: Day 1 up to Day 95
Population: Safety Analysis Set included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Number analyzed (Participants) | 23 | 23 | 25 | 27
percentage of participants
  Hematocrit <0.8 x LLN (n=22,23,25,27) | 0 | 0 | 0 | 0
  Hematocrit >1.2 x ULN (n=22,23,25,27) | 0 | 0 | 0 | 0
  Hemoglobin <0.8 x LLN (n=22,23,25,27) | 0 | 0 | 0 | 0
  Hemoglobin >1.2 x ULN (n=22,23,25,27) | 0 | 0 | 0 | 0
  Platelet Count <75 x 10^3/μL (n=22,23,25,27) | 0 | 0 | 0 | 0
  Platelet Count >600 x 10^3/μL (n=22,23,25,27) | 0 | 0 | 0 | 0
  Red Blood Cells <0.8 x LLN (n=22,23,25,27) | 0 | 0 | 0 | 0
  Red Blood Cells >1.2 x ULN (n=22,23,25,27) | 0 | 0 | 0 | 0
  White Blood Cells <0.5 x LLN (n=22,23,25,27) | 0 | 0 | 0 | 0
  White Blood Cells >1.5 x ULN (n=22,23,25,27) | 0 | 0 | 0 | 0
  Alanine Aminotransferase >3 x ULN | 0 | 0 | 0 | 0
  Albumin <2.5 g/dL | 0 | 0 | 0 | 0
  Alkaline Phosphatase >3 x ULN | 0 | 0 | 0 | 0
  Aspartate Aminotransferase >3xULN | 0 | 0 | 0 | 0
  Blood Urea Nitrogen >10.7 mmol/L | 0 | 0 | 0 | 0
  Calcium <1.75 mmol/L | 0 | 0 | 0 | 0
  Calcium >2.88 mmol/L | 0 | 0 | 0 | 0
  Creatine Kinase >5 x ULN | 0 | 0 | 0 | 0
  Creatinine >2.0 mg/dL | 0 | 0 | 0 | 0
  Gamma Glutamyl Transpeptidase >3xULN | 0 | 0 | 0 | 0
  Potassium <3.0 mmol/L | 0 | 0 | 0 | 0
  Potassium >6.0 mmol/L | 0 | 0 | 0 | 0
  Sodium <130 mmol/L | 0 | 0 | 0 | 0
  Sodium >150 mmol/L | 0 | 0 | 0 | 0
  Total Bilirubin >2.0 mg/dL | 0 | 0 | 0 | 0
  Total Protein <0.8 x LLN | 0 | 0 | 0 | 0
  Total Protein >1.2 x ULN | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants With Markedly Abnormal Vital Sign Measurements at Least Once Post-dose
Description: The percentage of participants who meet markedly abnormal criteria for vital signs, including oral body temperature, respiration rate, pulse, and resting blood pressure and after standing.
Time Frame: Day 1 up to Day 95
Population: Safety Analysis Set included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Number analyzed (Participants) | 23 | 23 | 25 | 27
percentage of participants
  Pulse <50 bpm | 26.1 | 21.7 | 28.0 | 33.3
  Pulse >120 bpm | 0 | 0 | 0 | 0
  Systolic Blood Pressure <85 mmHg | 0 | 0 | 0 | 0
  Systolic Blood Pressure >180 mmHg | 0 | 0 | 0 | 0
  Diastolic Blood Pressure <50 mmHg | 0 | 8.7 | 0 | 11.1
  Diastolic Blood Pressure >110 mmHg | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) Parameters at Least Once Post-Dose
Description: The percentage of participants who meet markedly abnormal criteria specified by the protocol and statistical analysis plan=abnormal clinically significant.
Time Frame: Day 1 up to Day 95
Population: Safety Analysis Set included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Number analyzed (Participants) | 23 | 23 | 25 | 27
percentage of participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (Up to ).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | A: Placebo | B: Donepezil 10 mg | C: Roflumilast Dose A | D: Roflumilast Dose A + Donepezil 10 mg
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/23 | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 7/23 | 9/23 | 5/25 | 12/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Placebo (N=23) | B: Donepezil 10 mg (N=23) | C: Roflumilast Dose A (N=25) | D: Roflumilast Dose A + Donepezil 10 mg (N=27)
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A: Placebo (N=23) | B: Donepezil 10 mg (N=23) | C: Roflumilast Dose A (N=25) | D: Roflumilast Dose A + Donepezil 10 mg (N=27)
Dizziness (Nervous system disorders) | 6 | 3 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 4 | 2 | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 5
Vision blurred (Eye disorders) | 1 | 3 | 2 | 2
Headache (Nervous system disorders) | 1 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.